CLINICAL TRIAL: NCT01621776
Title: Comparison of Effectiveness of Glulisine and Lispro in Decreasing Post-Prandial Hyperglycemia in a Real-World Setting
Brief Title: Effect of Apidra Compared to Humalog in Decreasing Post-Prandial Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3842011
Record Dates: First submitted 2012-06-11; First posted 2012-06-18 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-01

CONDITIONS: Type 1 Diabetes
Keywords: post-prandial hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Humalog (Active Comparator): Subjects on this treatment arm will receive Humalog insulin for their bolus doses, with doses optimized individually to achieve glycemic targets at daily medical rounds with their cabin physicians.
  Interventions: Drug: Humalog
- Apidra (Active Comparator): Subjects on this treatment arm will receive Apidra insulin for their bolus doses, with doses optimized individually to achieve glycemic targets at daily medical rounds with their cabin physicians.
  Interventions: Drug: Apidra
- Novolog (Active Comparator): Subjects on this treatment arm will receive Novolog insulin for their bolus doses, with doses optimized individually to achieve glycemic targets at daily medical rounds with their cabin physicians. (NOTE: This arm was only for one year of the study which was the 2012 camp session.)
  Interventions: Drug: Novolog

INTERVENTIONS:
Drug: Apidra — Subjects on this treatment arm will receive Apidra insulin for their bolus doses, with doses optimized individually to achieve glycemic targets at daily medical rounds with their cabin physicians.
  Other Names: Insulin glulisine
  Arms: Apidra
Drug: Humalog — Subjects on this treatment arm will receive Humalog insulin for their bolus doses, with doses optimized individually to achieve glycemic targets at daily medical rounds with their cabin physicians.
  Other Names: Insulin lispro
  Arms: Humalog
Drug: Novolog — Subjects on this treatment arm will receive Novolog insulin for their bolus doses, with doses optimized individually to achieve glycemic targets at daily medical rounds with their cabin physicians. (NOTE: This arm was only for one year of the study which was the 2012 camp session.)
  Other Names: Insulin aspart
  Arms: Novolog

SUMMARY:
This study aims to compare the post-meal blood glucose values of two drugs in a "real-world" setting.

DETAILED DESCRIPTION:
This is a randomized, open-label trial that aims to compare the glycemic excursion following food intake following post-meal injection of Glulisine (Apidra) insulin and Lispro (Humalog) insulin in a real-world setting. Children participating in the Florida Camp for Children and Youth with Diabetes will be randomized to receive either Glulisine or Apidra to cover carbohydrates after meals. The difference in blood glucose values will be analyzed before and 2 hours after meals to see if there is a difference in post-prandial hyperglycemia between groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 Diabetes
* Children and Youth attending Florida Diabetes Camp in DeLand, FL

Exclusion Criteria:

* only campers participating in sessions I and II are eligible to participate

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Silverstein, M.D., Principal Investigator — University of Florida
Locations (1):
- Camp Winona, DeLeon Springs, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the Florida Camp for Children & Youth with Diabetes during the summers of 2011 and 2012. In the summer of 2012 an additional arm was added to the study to include Novolog.
Pre-assignment Details: There were 107 participants consented to the study. 8 participants were withdrawn prior to randomization to the study.
Period: Overall Study
Arm/Group | Humalog | Apidra | Novolog
Started | 41 | 40 | 18
Completed | 41 | 40 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In the first year (Camp 2011) there were 2 arms, the Humalog and Apidra. In the second year (Camp 2012) there were 3 arms, the Humalog, Apidra, and Novolog. Therefore, there will be more participants in the Humalog and Apidra arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Humalog | Apidra | Novolog | Total
Number analyzed (Participants) | 41 | 40 | 18 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 40 | 18 | 99
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 11 | 53
  Male | 20 | 19 | 7 | 46
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 18 | 99

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between Pre- and 120 Minute Post-prandial Blood Glucose Concentrations at Lunch.
Description: Blood glucose concentrations were measured prior to and 90 minutes following lunch. Analysis was based on intention to treat. While missing data was imputed, it was known that this data was 'not missing at random' thus violating standard statistical assumptions with imputation. Therefore imputed data was not included in the final model.
  The number of participants for analysis was based upon a convenience sample of individuals attending Florida Camp for Children and Youth with Diabetes at Camp Winona.
Time Frame: averaged over 5 days
Population: Post-Prandial Blood Glucose Values [Within 90 minutes following the completion of participant lunch]
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Humalog | Apidra | Novolog
Number analyzed (Participants) | 41 | 40 | 18
mg/dl | 146.69 (79.19) | 143.68 (79.48) | 149.02 (71.56)
Statistical Analysis 1: Comparison: Humalog vs Apidra vs Novolog; Test type: Superiority or Other; p = .971, ANOVA; Mean Difference (Final Values) = 145.10, 95% CI [129.73 to 160.47], Standard Deviation 78.04 — This is a three arm study that is not seeking to engage in comparison between individual arms, therefore the mean difference across the study arms is reported

2. Secondary Outcome: Difference Between Pre- and 120 Minute Post-prandial Blood Glucose Concentrations at Dinner
Description: Blood glucose concentrations were measured prior to and 120 minutes following dinner. Analysis was based on intention to treat. While missing data was imputed, it was known that this data was 'not missing at random' thus violating standard statistical assumptions with imputation. Therefore imputed data was not included in the final model.
Time Frame: averaged over 5 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Humalog | Apidra | Novolog
Number analyzed (Participants) | 41 | 40 | 18
mg/dl | 170.57 (50.54) | 160.96 (73.54) | 153.46 (62.72)
Statistical Analysis 1: Comparison: Humalog vs Apidra vs Novolog; Test type: Superiority or Other; p = .698, ANOVA; Mean Difference (Final Values) = 161.09, 95% CI 2-sided [144.91 to 177.28], Standard Deviation 62.67 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Difference Between Pre- and 120 Minute Post-prandial Blood Glucose Concentrations at Breakfast
Description: Blood glucose concentrations were measured prior to and 120 minutes following breakfast. Analysis was based on intention to treat. While missing data was imputed, it was known that this data was 'not missing at random' thus violating standard statistical assumptions with imputation. Therefore imputed data was not included in the final model.
Time Frame: averaged over 5 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Humalog | Apidra | Novolog
Number analyzed (Participants) | 41 | 40 | 18
mg/dl | 225.62 (111.48) | 225.46 (81.14) | 208.64 (76.53)
Statistical Analysis 1: Comparison: Humalog vs Apidra vs Novolog; Test type: Superiority or Other; p = .806, ANOVA; Mean Difference (Final Values) = 220.46, 95% CI 2-sided [197.22 to 243.71], Standard Deviation 89.97 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: July 2011 through July 2012
Arm/Group | Humalog | Apidra | Novolog
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/18
Other Adverse Events (participants affected / at risk) | 41/41 | 40/40 | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog (N=41) | Apidra (N=40) | Novolog (N=18)
Hypoglycemic Event (Endocrine disorders) | 41 (105) | 40 (124) | 18 (35) — The participants have a diagnosis of diabetes. A hypoglycemic event is not an unusual occurrence for them to experience.

LIMITATIONS AND CAVEATS:
In the first year (Camp 2011) there were 2 arms, the Humalog and Apidra. In the second year (Camp 2012) there were 3 arms, the Humalog, Apidra, and Novolog. Therefore, there will be more participants in the Humalog and Apidra arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No